CLINICAL TRIAL: NCT05786248
Title: MOdification of Fluid Distribution in 90 Minutes : Pilot Study - MORFE 90
Brief Title: MOdification of Fluid Distribution in 90 Minutes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MORFE90
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea; Fluid Retention
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Impedancemtry (Other): measurement of fluid shift by impedancemetry, recording by polysomnography, measurement of neck, calf and ankle perimeters, at different times: 0 min (T0), 30min (T30), 90min (T90), and the next day on waking
  Interventions: Other: Impedancemetry

INTERVENTIONS:
Other: Impedancemetry — the impedance measurement electrodes are placed on the lower limbs and neck. After the first measurement, the patients are invited to lie down. A new series of measurements will be performed at 30 (T30), 90 minutes (T90) and in the morning.

SUMMARY:
Obstructive Sleep Apnea-Hypopnea Syndrome (OSAHS) is a cardiovascular risk factor due to intermittent hypoxia phenomena. Several etiological factors are involved in the pathogenesis of OSAS. Among them, the rostro-caudal displacement of fluid during dorsal decubitus has been highlighted. Under the effect of gravity, an accumulation of fluid is possible in the lower limbs, redistributing itself towards the upper parts of the body during the supine position.

This phenomenon of fluid shift is usually evaluated by impedancemetry after a night in the supine position. However, some authors have shown that fluid shift occurs within 90 minutes after supine. Thus, in the perspective of future studies, in order to simplify the implementation of this evaluation and to reduce the time of hospitalization necessary for the subjects participating in the study, we would like to verify the correlation between the impedancemetry measurement at T 90 min and that obtained after one night of supine position. This is a single-center, prospective, open-label study at the Poitiers University Hospital. We will include 30 patients over 18 years of age admitted to the regional sleep pathology center for suspected nocturnal respiratory disorders to receive polysomnography and able to provide written consent.We excluded : patients younger than 18 years of age, A history of vascular surgery of the lower limbs such as varicose vein surgery, vascular bypass surgery, carcinological surgery with lymph node dissection, the presence of metallic implants in the lower limbs or spine or implantable cardiac devices, those not receiving Social Securitý or not receiving it through a third party, persons receiving enhanced protection, namely minors, and persons deprived of libertý by a judicial or administrative decision, persons staying in a health or social institution, and adults under legal protection.we will perform an impedance measurement at T0, T30, T90, and after overnight supine. Impedance measurement is performed using electrodes delivering a low intensity current of known frequency allowing the study of the liquid volume.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients requiring polysomnography at the regional sleep pathology center for suspected nocturnal breathing disorders
* Patients able to give their non-opposition

Exclusion Criteria:

* The presence of metallic implants in the lower limbs or spine or implantable pacemakers because of possible interference with the impedance signals
* A history of amputation of both lower limbs
* Persons benefiting from reinforced protection, namely minors, persons deprived of libertý by a judicial or administrative decision, persons staying in a health or social institution and adults under legal protection, persons in emergency situations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
To evaluate the agreement between impedancemetry measurements at T90 minutes and impedancemetry measurements after an overnight supine position in the assessment of Fluid-Shift. | 90 minutes
  The criterion evaluated is the fluid volume redistributed between the lower limbs and the neck by impedancemetry between T0 and T90 minutes and between T0 and after one night of supine.The concordance criterion is the intraclass correlation coefficient (ICC).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No